CLINICAL TRIAL: NCT05362214
Title: Effects of Different Guiding Strategies on Biomechanics of Human Movement.
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Fong Chin Su, Distinguished Professor, National Cheng-Kung University Hospital
Other Study IDs: 109-423
Record Dates: First submitted 2022-04-14; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Healthy Aging
Keywords: Baduanjin Qigong; Visual and Auditory Cues; Center of Pressure (COP); Smoothness of Arm Movement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Audio (no visual cue): The condition that a participant has to perform Baduanjin exercise by following the audio guidance/illustration according to the reference of Baduanjin practicing video.
- Video (2D visual cue): The condition that a participant has to perform Baduanjin exercise by following the video guidance/illustration according to the reference of Baduanjin practicing video.
- Drone (3D visual cue): The condition that a participant has to perform Baduanjin exercise by following the drone guiding system including a guidance from drone and audio illustration regarding the reference of Baduanjin practicing video.

SUMMARY:
With regards to the increase in the aging population globally, how to build up a successfully aging society has become the main issue in health care and socioeconomic. In addition, living with high physical function is one of the main goals and solutions, and exercising regularly is a direct and obvious way to achieve this goal. However, being elderly, it might not be easy for them to practice or do exercise every day due to some of their limitations such as learning difficulty and lack of motivation.

Nowadays, there are many different types of exercise supporting tools, which are in terms of visual or auditory cues, including two-dimensional (2D) or three-dimensional (3D) cues. Accordingly, several studies mentioned the positive outcomes of using a 3D visual cue compared with using the 2D one. Also, a study found that combining visual and auditory cues together resulted in a better perception than using either one alone.

Coupled with a coming of a small flyable robot so-called "drone", which can be programmed to fly autonomously in a 3D space, a few research teams applied it in many interactive applications with humans such as sports education relating for example dancing and boxing. Moreover, there was a research team that explored the interaction between a human and a drone in a close-range design by controlling the drone using both hands movement, which was inspired by Tai Chi martial art exercise. As a result, they found important findings of the calming and focusing experience of the participants due to the low level of constant propeller noise of the drone.

Regarding this, the investigators assumed that applying a drone, which can be recognized as a 3D visual cue, to a kind of exercise may provide some benefits in terms of physical health. In addition, the investigators applied it to a simple Chinese martial art exercise called "Baduanjin Qigong" since it was recommended for everyone, especially for the elderly because of its low requirement for physical and cognitive abilities.

However, based on our findings, there is no published information about the effects of the drone as a visual cue or exercise guiding tool in terms of biomechanical effects of human motion. Therefore, these effects would be observed throughout this study.

Besides, the investigators hypothesized that exercising with the drone, which is a 3D visual cue in this study, could provide a significant difference in biomechanics effects such as the center of pressure (COP) and smoothness of the arm when compared with using a 2D visual cue like video, or no visual cue like the audio illustration. Also, resulting in a positive direction as an exercise guiding tool for the elderly such as increasing their motivation during exercise.

ELIGIBILITY:
Inclusion Criteria:

* 20 years old above
* Able to perform regular exercise
* Able to understand Chinese or Taiwanese language
* Never practice Baduanjin Qigong

Exclusion Criteria:

* Having illness or diseases that cannot perform physical exercise such as musculoskeletal disease.
* Having any kinds of chronic disease that might be more activated by performing Baduanjin exercise such as cardiovascular diseases, chronic respiratory diseases, osteoporosis, etc.
* Having chronic diseases that cannot perform Baduanjin exercise according to the experimental protocols such as blindness, deafness and hearing impairment, or Alzheimer's diseases, etc.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of Tainan city, Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Center of pressure (COP) | 2 hours
  The center of pressure (COP) of every participant while performing each selected movement of Baduanjin exercise were observed with regards to the three different guiding strategies including audio, video, and drone.
Smoothness of arm movement | 2 hours
  The smoothness of arm movement of every participant while performing each selected movement of Baduanjin exercise were observed with regards to the three different guiding strategies including audio, video, and drone.
Motivation and feedback of participants toward the drone guiding system | 2 hour
  Motivation and feedback of the participants toward the drone guiding system were measured through a questionnaire using Agree Disagree Rating Questions (5 scales: strongly agree, agree, neither agree nor disagree(normal), disagree, strongly disagree).

SECONDARY OUTCOMES:
Accuracy of the drone guiding system | 2 hours
  The accuracy of the drone guiding system was evaluated according to the paths that the drone could perform compared with the preprogrammed paths for each selected movement of Baduanjin exercise. However, only the endpoints of the drone were evaluated for accuracy testing since the inputs of the preprogrammed paths were specific endpoint values, not the entire trajectories of the drone.
Precision of the drone guiding system | 2 hours
  The precision of the drone guiding system was evaluated according to the entire trajectories that the drone performed in the 2nd, 3rd, 4th, and 5th times compared with the trajectory that the drone performed in the 1st time.

CONTACTS AND LOCATIONS:
Overall Officials: Fong-Chin Su, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
The study is still under the patent filling process.

REFERENCES:
- [Background] Lin PS, Hsieh CC, Cheng HS, Tseng TJ, Su SC. Association between Physical Fitness and Successful Aging in Taiwanese Older Adults. PLoS One. 2016 Mar 10;11(3):e0150389. doi: 10.1371/journal.pone.0150389. eCollection 2016. PMID 26963614
- [Background] McPhee JS, French DP, Jackson D, Nazroo J, Pendleton N, Degens H. Physical activity in older age: perspectives for healthy ageing and frailty. Biogerontology. 2016 Jun;17(3):567-80. doi: 10.1007/s10522-016-9641-0. Epub 2016 Mar 2. PMID 26936444
- [Background] Zou L, SasaKi JE, Wang H, Xiao Z, Fang Q, Zhang M. A Systematic Review and Meta-Analysis Baduanjin Qigong for Health Benefits: Randomized Controlled Trials. Evid Based Complement Alternat Med. 2017;2017:4548706. doi: 10.1155/2017/4548706. Epub 2017 Mar 7. PMID 28367223
- [Background] Liu XY, Gao J, Yin BX, Yang XY, Bai DX. Efficacy of Ba Duan Jin in Improving Balance: A Study in Chinese Community-Dwelling Older Adults. J Gerontol Nurs. 2016 May 1;42(5):38-46. doi: 10.3928/00989134-20160201-03. PMID 27110739
- [Background] Zheng G, Fang Q, Chen B, Yi H, Lin Q, Chen L. Qualitative Evaluation of Baduanjin (Traditional Chinese Qigong) on Health Promotion among an Elderly Community Population at Risk for Ischemic Stroke. Evid Based Complement Alternat Med. 2015;2015:893215. doi: 10.1155/2015/893215. Epub 2015 Sep 21. PMID 26483845
- [Background] Tse CK, Yu CK. The Effects of Visual Cues, Blindfolding, Synesthetic Experience, and Musical Training on Pure-Tone Frequency Discrimination. Behav Sci (Basel). 2018 Dec 24;9(1):2. doi: 10.3390/bs9010002. PMID 30586857
- [Background] Pierno AC, Caria A, Castiello U. Comparing effects of 2-D and 3-D visual cues during aurally aided target acquisition. Hum Factors. 2004 Winter;46(4):728-37. doi: 10.1518/hfes.46.4.728.56815. PMID 15709333
- [Background] Sodhi R, Benko H, Wilson A. LightGuide. Proceedings of the SIGCHI Conference on Human Factors in Computing Systems. 2012 May 5;179-188. doi: 10.1145/2207676.2207702.
- [Background] La Delfa J, Baytas MA, Patibanda R, Ngari H, Khot RA, Mueller F'F. Drone Chi: Somaesthetic human-drone interaction. Proceedings of the 2020 CHI Conference on Human Factors in Computing Systems. 2020 April 23;1-13. doi: 10.1145/3313831.3376786.
- [Background] Kim H, Landay JA. Aeroquake: Drone Augmented Dance. Proceedings of the 2018 Designing Interactive Systems Conference. 2018 June 8;691-701. doi: 10.1145/3196709.3196798.
- [Background] Eriksson S, Unander-Scharin Å, Trichon V, Unander-Scharin C, Kjellström H, Höök K. Dancing with drones: Crafting Novel Artistic Expressions Through Intercorporeality. Proceedings of the 2019 CHI Conference on Human Factors in Computing Systems. 2019 May 2;1-12. doi: 10.1145/3290605.3300847.
- [Background] Zwaan SG, Barakova EI. Boxing against Drones: Drones in Sports Education. Proceedings of the The 15th International Conference on Interaction Design and Children. 2016 June 21;607-612. doi: 10.1145/2930674.2935991.